CLINICAL TRIAL: NCT07304661
Title: Comparison of Pulse Pressure Variation and LVOT VTI-Based Cardiac Output Changes During Passive Leg Raising Maneuver in Predicting Fluid Responsiveness in Mechanically Ventilated Critically Ill Patients: A Prospective Observational Study
Brief Title: Comparison of PPV and LVOT VTI During Passive Leg Raising to Predict Fluid Responsiveness
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ahmet Salih Tüzen, MD, Medical Doctor, Izmir Katip Celebi University
Other Study IDs: 2025-SAEK-0811
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hemodynamic Instability; Hypovolemia; Critical Illness; Pulse Pressure Variation
Keywords: Fluid Responsiveness; Passive Leg Raising; Pulse Pressure Variation; LVOT VTI; Cardiac Output; Echocardiography
MeSH Terms: conditions — Hypovolemia; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fluid Responders: Defined as an increase in LVOT VTI-based Cardiac Output (CO) of ≥ 10% from baseline.
- Fluid Non-Responders: Defined as an increase in LVOT VTI-based Cardiac Output (CO) of < 10% from baseline.

SUMMARY:
Hemodynamic instability remains one of the leading causes of morbidity and mortality among critically ill patients in intensive care units. One major contributor to this instability is intravascular fluid deficit. Although fluid administration is often preferred as an initial intervention, inaccurate estimation of fluid requirements carries significant risks. Inadequate resuscitation may lead to tissue hypoperfusion and organ dysfunction, whereas excessive fluid loading is associated with pulmonary edema, increased intra-abdominal pressure, multi-organ dysfunction, and increased mortality. Consequently, reliable prediction of fluid responsiveness is considered a critical determinant in modern intensive care management.

The limited reliability of static parameters in predicting fluid responsiveness and the fact that PPV retains its validity only under specific clinical conditions highlight the need for more effective methods. In recent years, hemodynamic changes assessed during the passive leg raising (PLR) maneuver have gained prominence; particularly, left ventricular outflow tract velocity time integral (LVOT VTI)-based cardiac output measurements have been identified as a strong parameter for predicting fluid responsiveness . Moreover, changes in pulse pressure variation (PPV) during PLR have also been reported as a potential predictor; however, the number of studies prospectively comparing PPV variation and LVOT VTI-based cardiac output change within the same patient population remains limited . Therefore, the proposed study aims to fill this gap in the literature and contribute to fluid management in the intensive care setting.

The aim of this study is to compare the performance of PPV variation and LVOT VTI-based cardiac output change after the PLR maneuver in predicting fluid responsiveness among mechanically ventilated critically ill patients, and to determine the diagnostic value of both methods. The findings of the present study are expected to support more reliable decision-making in fluid therapy and provide clinical evidence toward the individualization of fluid management in intensive care practice.

DETAILED DESCRIPTION:
This study is designed as a prospective observational trial. No additional intervention, procedure, or treatment beyond standard clinical practice will be performed. All data will be obtained during routine clinical management in our intensive care unit.

In mechanically ventilated patients with suspected fluid deficit, the passive leg raising (PLR) maneuver is applied as part of standard practice, during which changes in pulse pressure variation (PPV) are recorded by invasive arterial monitoring.

In this observational study, transthoracic echocardiographic (TTE) measurements of LVOT VTI will be performed by an experienced operator in addition to routine practice. Using pulse wave Doppler (PW), LVOT VTI will be recorded, and stroke volume (SV) and cardiac output (CO) will be calculated by multiplying the LVOT VTI value by the LVOT diameter. Consequently, changes in PPV and LVOT VTI-based CO during PLR will be compared.

Following TTE measurements of LVOT VTI and LVOT diameter in both the semi-recumbent position (45°) and immediately after PLR, SV and CO will be calculated. Based on these measurements, patients will be allocated into two groups:

* Fluid responsive: Patients showing ≥10% increase in LVOT VTI-based CO following PLR
* Non-fluid responsive: Patients showing <10% change in LVOT VTI-based CO following PLR

After grouping patients accordingly, PPV changes during PLR will be compared between the two groups. This will allow evaluation of the predictive performance of PPV variation relative to LVOT VTI-based CO change in determining fluid responsiveness. All measurements will be performed by an experienced clinician without disrupting standard patient care. No additional fluid loading, invasive procedures, or therapeutic interventions will be undertaken throughout the study.

The primary aim is to compare the diagnostic performance of PPV variation and LVOT VTI-based cardiac output changes following a PLR maneuver in predicting fluid responsiveness. The study seeks to determine the diagnostic value of both methods to support more individualised fluid management.

The recorded data will include:

* Pre- and post-PLR LVOT VTI, stroke volume, cardiac output, and PPV values
* Routine monitoring parameters (systolic/diastolic blood pressure, mean arterial pressure, heart rate, and SpO₂)
* Demographic characteristics (age, sex, comorbidities) retrieved through the hospital database

Informed consent will be obtained from all participating patients or their legally authorized representatives.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥18 years
2. Patients admitted to the intensive care unit receiving mechanical ventilation
3. Presence of suspected intravascular fluid deficit (hypotension, negative fluid balance, or clinical signs of peripheral hypoperfusion)
4. Patients in sinus rhythm
5. Presence of invasive arterial blood pressure monitoring
6. Adequate echocardiographic window allowing transthoracic echocardiographic measurement of LVOT VTI
7. Patients ventilated with tidal volume ≥8 mL/kg (ideal body weight)
8. Hemodynamically stable enough to allow measurement

Exclusion Criteria:

1. Patients under 18 years of age
2. Presence of atrial fibrillation or significant arrhythmias such as frequent ventricular or atrial ectopy
3. Severe right ventricular dysfunction or significant tricuspid regurgitation
4. Advanced aortic valve disease (severe stenosis or severe regurgitation)
5. Patients with significant spontaneous breathing effort
6. Patients receiving lung-protective low tidal volume ventilation strategy (<8 mL/kg) due to ARDS
7. Inadequate echocardiographic window for LVOT VTI assessment
8. Severe hemodynamic instability during measurement (sudden vasopressor escalation or need for resuscitation)
9. Patients who refuse to participate or from whom written informed consent cannot be obtained from themselves or a first-degree relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult critically ill patients admitted to the Intensive Care Unit (ICU) who are receiving mechanical ventilation support. Eligible participants are those identified by the intensive care team as having a suspected intravascular fluid deficit, for whom a fluid responsiveness assessment is clinically indicated. The cohort specifically targets patients undergoing the Passive Leg Raising (PLR) maneuver as part of routine standard practice, where invasive arterial monitoring is available to record Pulse Pressure Variation (PPV).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pulse Pressure Variation (Delta PPV) | Baseline (T0) and between 60 seconds after the PLR maneuver.
  Pulse Pressure Variation (PPV) is recorded via invasive arterial monitoring at baseline (T0, semi-sitting) and during the Passive Leg Raising maneuver (T1).

SECONDARY OUTCOMES:
Percentage Change in Cardiac Output (Delta CO) | Baseline (T0) and between 60 seconds after the PLR maneuver.
  Cardiac Output (CO) is calculated using the Left Ventricular Outflow Tract Velocity Time Integral (LVOT VTI) and the LVOT diameter measured via transthoracic echocardiography.
Correlation between Delta PPV and Delta CO | Baseline (T0) and between 60 seconds after the PLR maneuver.
  Correlation Coefficient (r) between PPV Change and Cardiac Output Change
Hemodynamic Parameter Changes (MAP, HR) | Baseline (T0) and between 60 seconds after the PLR maneuver.
  Measurement of changes in mean arterial pressure and heart rate before and after PLR and comparison between groups.
Diagnostic Accuracy (ROC-AUC, Sensitivity, Specificity, Cut-off) | Baseline (T0) and between 60 seconds after the PLR maneuver.
  Evaluation of diagnostic performance of ΔPPV and ΔCO using receiver operating characteristic (ROC) analysis, including AUC, optimal cut-off value, sensitivity, and specificity for predicting fluid responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Aksun, Principal Investigator — Izmir Katip Celebi University Atatürk Training and Research Hospital
Locations (1):
- Izmir Katip Celebi University Atatürk Training and Research Hospital İzmir, , Turkey, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All data necessary to support the study protocol, including de-identified individual participant data (IPD) related to study protocol, and primary and secondary outcome measures, will be made available upon reasonable request from qualified researchers for academic purposes, in accordance with institutional and ethical guidelines.